CLINICAL TRIAL: NCT01495468
Title: Pegylated Somatropin in the Treatment of Children With Growth Hormone Deficient：A Multicenter, Randomized, Open-label, Controlled Phase Ⅲ Clinical Trial
Brief Title: Phase III Clinical Study of Pegylated Somatropin (PEG Somatropin) to Treat Growth Hormone Deficiency Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Capital Medical University (Other); Children's Hospital of Fudan University (Other); The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci-004-CT
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2011-12

CONDITIONS: Growth Hormone Deficiency
Keywords: pegylated somatropin; PEG-rhGH; growth hormone; Growth Hormone Deficiency; phase III study
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: PEG-somatropin — drug:pegylated somatropin 0.2mg/(kg.w), once per week for 6 months drug: Jintropin AQ, 0.25mg/(kg.w), once per day for 6 months
  Other Names: recombinant human growth hormone; peglyated growth hormone; PEG-GH

SUMMARY:
This was a multicenter, randomized, open-label, parallel controlled phase III study, compared pegylated somatropin with Jintropin AQ (somatropin liquid injection, daily administration formulation).

All the subjects were randomized into two groups, test group (PEG somatorpin) and control group (Jintropin AQ), 200 children were enrolled in test group and 100 children were enrolled in control group. Considering the case loss during the clinical study, 20% of the patients were added in each of the group, that is 240 children were in test group and 120 children were in control group, totally 360 children were enrolled in the phase III clinical study.

Whole treatment were lasted for 6 months, 4 times of follow-up were carried out at the point of baseline, 1 month, 3 month and 6 month after treatment. The evaluation of the primary time point was 3 month and 6 month after treatment, if the treatment was less than 6 months, the evaluation would be made when the treatment is finished.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects have a height less than two standard deviations (SD) below the median height for individuals of he same age or height,the growth velocity (CV≤4.0 cm/yr),GH peak concentration <7.0ng/ml in two difference provocative tests, Bone age (BA) ≤9 years in girls and ≤10 years in boys, at least 2 year less than his/her chronological age (CA)
* be in preadolescence (Tanner stage 1) and have a CA > 3 years
* have a height value recorded 3 months before the start of GH treatment to calculate pre-treatment GV.
* receive no prior GH treatment.
* sign informed consent

Exclusion Criteria:

* 1. patients positive for hepatitis B e-antibody (HBeAb), hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg)
* 2.Known hypersensitivity to Somatropin or any other components of the study product.
* 3. severe cardiopulmonary or hematological diseases, a current or past history of malignant tumors, immunodeficiency diseases, or mental diseases
* 4. with other growth disorders, such as Turner syndrome, constitutional delay of growth and puberty, and Laron syndrome
* 5. Subjects took part in other clinical trial study during 3 months.
* 6. Other conditions which in the opinion of the investigator preclude enrollment into the study.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 343 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
yearly growth velocity | 6 months
  growth velocity add as GV was the primary outcome measure

SECONDARY OUTCOMES:
Ht SDSca | 6 months
  Ht SDSca was calculated by dividing the difference between the actual height of a patient and the mean height of the population for that chronological age by the standard deviation (SD) of the height of the population for that chronological age
IGF-l | 6 months
IGFBP-3 | 6 months
bone maturity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, Ph. D, Principal Investigator — Tongji Hospital
Locations (6):
- China (6):
  - Beijing
  - Changchun
  - Guangzhou
  - Hangzhou
  - Shanghai
  - Wuhan

REFERENCES:
- [Result] Luo X, Hou L, Liang L, Dong G, Shen S, Zhao Z, Gong CX, Li Y, Du ML, Su Z, Du H, Yan C. Long-acting PEGylated recombinant human growth hormone (Jintrolong) for children with growth hormone deficiency: phase II and phase III multicenter, randomized studies. Eur J Endocrinol. 2017 Aug;177(2):195-205. doi: 10.1530/EJE-16-0905. Epub 2017 May 31. PMID 28566441